CLINICAL TRIAL: NCT00363896
Title: Clinical Trial Assessing Efficacy and Safety of LAS34273 in Moderate to Severe Stable Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: A Trial Assessing LAS34273 in Moderate to Severe Stable Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M/34273/30; ACCLAIM I (Other: Almirall,S.A.); CT000740 (Other: Almirall,S.A.)
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2012-11-01 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Lung function; Exacerbations; Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aclidinium 200 μg once-daily (Experimental): Aclidinium bromide 200 μg once-daily by inhalation
  Interventions: Drug: Aclidinium bromide
- Placebo (Placebo Comparator): Placebo once-daily via inhalation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium bromide — Aclidinium bromide 200 μg once-daily via inhalation via the Eklira Genuair® inhaler: 1 puff in the morning for 52 weeks
  Arms: Aclidinium 200 μg once-daily
Drug: Placebo — Placebo once-daily via inhalation: 1 puff in the morning for 52 weeks
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of LAS 34273 compared to placebo in patients with moderate to severe COPD during one year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥ 40 years with a clinical diagnosis of moderate to severe stable COPD

Exclusion Criteria:

* History or current diagnosis of asthma, recent respiratory tract infection or acute COPD exacerbation, life expectancy of less than 1 year, known symptomatic prostatic hypertrophy, bladder neck obstruction or narrow-angle glaucoma

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 843 (Actual)
Dates: Start 2006-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (132):
- Almirall Investigational Sites#947, Les Escaldes, Andorra
- Austria (5):
  - Almirall Investigational Sites#645, Graz
  - Almirall Investigational Sites#646, Innsbruck
  - Almirall Investigational Sites#644, Linz
  - Almirall Investigational Sites#647, Vienna
  - Almirall Investigational Sites#649, Vienna
- Belgium (4):
  - Almirall Investigational Sites#110, Aalst
  - Almirall Investigational Sites#394, Brussels
  - Almirall Investigational Sites#651, Edegem
  - Almirall Investigational Sites#393, Namur
- Bulgaria (10):
  - Almirall Investigational Sites#658, Burgas
  - Almirall Investigational Sites#653, Pleven
  - Almirall Investigational Sites#654, Plovdiv
  - Almirall Investigational Sites#656, Rousse
  - Almirall Investigational Sites#652, Sofia
  - Almirall Investigational Sites#657, Sofia
  - Almirall Investigational Sites#972, Sofia
  - Almirall Investigational Sites#971, Sofia
  - Almirall Investigational Sites#655, Varna
  - Almirall Investigational Sites#953, Veliko Tarnovo
- Czechia (8):
  - Almirall Investigational Sites#664, Lovosice
  - Almirall Investigational Sites#660, Neratovice
  - Almirall Investigational Sites#662, Pilsen
  - Almirall Investigational Sites#666, Prague
  - Almirall Investigational Sites#661, Prague
  - Almirall Investigational Sites#665, Tábor
  - Almirall Investigational Sites#659, Třemošná
  - Almirall Investigational Sites#954, Žatec
- Denmark (3):
  - Almirall Investigational Sites#398, Aalborg
  - Almirall Investigational Sites#390, Århus C
  - Almirall Investigational Sites#397, Odense C
- France (9):
  - Almirall Investigational Sites#594, Beuvry
  - Almirall Investigational Sites#593, Brest
  - Almirall Investigational Sites#750, Grasse
  - Almirall Investigational Sites#669, Montpellier
  - Almirall Investigational Sites#672, Paris
  - Almirall Investigational Sites#948, Perpignan
  - Almirall Investigational Sites#549, Rouen
  - Almirall Investigational Sites#671, Strasbourg
  - Almirall Investigational Sites#752, Vieux-Condé
- Germany (10):
  - Almirall Investigational Sites#678, Bad Wörishofen
  - Almirall Investigational Sites#758, Berlin
  - Almirall Investigational Sites#765, Berlin
  - Almirall Investigational Sites#680, Berlin
  - Almirall Investigational Sites#677, Berlin-Spandau
  - Almirall Investigational Sites#681, Bonn
  - Almirall Investigational Sites#191, Großhansdorf
  - Almirall Investigational Sites#766, Hamburg
  - Almirall Investigational Sites#757, Jena
  - Almirall Investigational Sites#675, Mainz
- Hungary (8):
  - Almirall Investigational Sites#684, Budapest
  - Almirall Investigational Sites#687, Debrecen
  - Almirall Investigational Sites#683, Debrecen
  - Almirall Investigational Sites#688, Nyíregyháza
  - Almirall Investigational Sites#686, Székesfehérvár
  - Almirall Investigational Sites#689, Szombathely
  - Almirall Investigational Sites#682, Tatabánya
  - Almirall Investigational Sites#685, Törökbálint
- Italy (6):
  - Almirall Investigational Sites#459, Genova
  - Almirall Investigational Sites#774, Milan
  - Almirall Investigational Sites#286, Modena
  - Almirall Investigational Sites#694, Napoli
  - Almirall Investigational Sites#635, Perugia
  - Almirall Investigational Sites#777, Pordenone
- Netherlands (4):
  - Almirall Investigational Sites#346, Breda
  - Almirall Investigational Sites#551, Eindhoven
  - Almirall Investigational Sites#348, Hengelo
  - Almirall Investigational Sites#695, Hoofddorp
- Poland (9):
  - Almirall Investigational Sites#700, Lodz
  - Almirall Investigational Sites#698, Lodz
  - Almirall Investigational Sites#697, Torun
  - Almirall Investigational Sites#699, Warsaw
  - Almirall Investigational Sites#696, Warsaw
  - Almirall Investigational Sites#702, Warsaw
  - Almirall Investigational Sites#706, Wroclaw
  - Almirall Investigational Sites#705, Zabrze
  - Almirall Investigational Sites#701, Zawadzkie
- Romania (9):
  - Almirall Investigational Sites#962, Brasov
  - Almirall Investigational Sites#970, Bucharest
  - Almirall Investigational Sites#714, Bucharest
  - Almirall Investigational Sites#713, Cluj-Napoca
  - Almirall Investigational Sites#712, Iași
  - Almirall Investigational Sites#961, Judetul Brasov
  - Almirall Investigational Sites#709, Palazu Mare
  - Almirall Investigational Sites#711, Târgu Mureş
  - Almirall Investigational Sites#715, Timișoara
- Russia (25):
  - Almirall Investigational Sites#462, Moscow
  - Almirall Investigational Sites#977, Moscow
  - Almirall Investigational Sites#721, Moscow
  - Almirall Investigational Sites#540, Moscow
  - Almirall Investigational Sites#967, Moscow
  - Almirall Investigational Sites#716, Moscow
  - Almirall Investigational Sites#722, Moscow
  - Almirall Investigational Sites#719, Moscow
  - Almirall Investigational Sites#582, Moscow
  - Almirall Investigational Sites#785, Moscow
  - Almirall Investigational Sites#976, Moscow
  - Almirall Investigational Sites#717, Moscow Region
  - Almirall Investigational Sites#588, Saint Petersburg
  - Almirall Investigational Sites#720, Saint Petersburg
  - Almirall Investigational Sites#965, Saint Petersburg
  - Almirall Investigational Sites#969, Saint Petersburg
  - Almirall Investigational Sites#543, Saint Petersburg
  - Almirall Investigational Sites#787, Saint Petersburg
  - Almirall Investigational Sites#975, Saint Petersburg
  - Almirall Investigational Sites#465, Saint Petersburg
  - Almirall Investigational Sites#966, Saint Petersburg
  - Almirall Investigational Sites#972, Saint Petersburg
  - Almirall Investigational Sites#786, Saint Petersburg
  - Almirall Investigational Sites#963, Saint Petersburg
  - Almirall Investigational Sites#718, Sochi
- Spain (8):
  - Almirall Investigational Sites#16, Badalona
  - Almirall Investigational Sites#7, Barcelona
  - Almirall Investigational Sites#317, Barcelona
  - Almirall Investigational Sites#61, Madrid
  - Almirall Investigational Sites#938, Málaga
  - Almirall Investigational Sites#727, Palma de Mallorca
  - Almirall Investigational Sites#723, Sant Joan d'Alacant
  - Almirall Investigational Sites#725, Terrassa
- United Kingdom (13):
  - Almirall Investigational Sites#738, Bedford
  - Almirall Investigational Sites#42, Bristol
  - Almirall Investigational Sites#734, Cottingham
  - Almirall Investigational Sites#735, Doncaster
  - Almirall Investigational Sites#788, Exeter
  - Almirall Investigational Sites#737, Hereford
  - Almirall Investigational Sites#784, London
  - Almirall Investigational Sites#37, London
  - Almirall Investigational Sites#730, Newcastle upon Tyne
  - Almirall Investigational Sites#731, Peterborough
  - Almirall Investigational Sites#728, Solihull
  - Almirall Investigational Sites#732, Suffolk
  - Almirall Investigational Sites#736, Windsor

REFERENCES:
- [Derived] Jones PW, Rennard SI, Agusti A, Chanez P, Magnussen H, Fabbri L, Donohue JF, Bateman ED, Gross NJ, Lamarca R, Caracta C, Gil EG. Efficacy and safety of once-daily aclidinium in chronic obstructive pulmonary disease. Respir Res. 2011 Apr 26;12(1):55. doi: 10.1186/1465-9921-12-55. PMID 21518460
- See also: Sponsor web site — http://www.almirall.com/webcorp2/cda/ImD_04_02.jsp
- See also: Co-Sponsor web site — http://www.frx.com/
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4056&filename=Synopsis_m-34273-30.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 132 sites: 1 in Andorra, 5 in Austria, 4 in Belgium, 10 in Bulgaria, 8 in the Czech Republic, 3 in Denmark, 9 in France, 10 in Germany, 8 in Hungary, 6 in Italy, 4 in Netherlands, 9 in Poland, 9 in Romania, 25 in Russia, 8 in Spain, 13 in the UK. First patient was screened in Aug 2006 and last patient visit was May 2008.
Pre-assignment Details: Following a screening visit, patients entered a 14-day run-in period during which they used inhaled salbutamol administered via a pressurised metered dose inhaler (pMDI) as rescue medication on an "as needed" basis. The 14-day run-in period was used to assess the stability of each patient's disease and baseline characteristics.
Groups:
- Aclidinium Bromide 200 μg Once-daily: Aclidinium bromide 200 μg once-daily by inhalation
- Placebo: Placebo by inhalation
Period: Overall Study
Arm/Group | Aclidinium Bromide 200 μg Once-daily | Placebo
Started | 627 | 216
Completed | 538 | 169
Not Completed | 89 | 47
Not completed — Withdrawal by Subject | 29 | 16
Not completed — Adverse Event | 24 | 13
Not completed — COPD exacerbation | 13 | 7
Not completed — Lack of Efficacy | 12 | 8
Not completed — Protocol Violation | 6 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Non-fulfilment of entry criteria | 1 | 0
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium Bromide 200 μg Once-daily | Placebo | Total
Number analyzed (Participants) | 627 | 216 | 843
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 378 | 134 | 512
  >=65 years | 249 | 82 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (8.2) | 61.9 (8.3) | 62.4 (8.2)
Gender [Count of Participants; unit: Participants]
  Female | 139 | 41 | 180
  Male | 488 | 175 | 663
Region of Enrollment [Number; unit: participants]
  Andorra | 3 | 1 | 4
  Austria | 14 | 4 | 18
  Belgium | 9 | 2 | 11
  Bulgaria | 61 | 20 | 81
  Czech Republic | 43 | 15 | 58
  Germany | 56 | 18 | 74
  Denmark | 9 | 3 | 12
  Spain | 31 | 10 | 41
  France | 36 | 14 | 50
  United Kingdom | 46 | 13 | 59
  Hungary | 39 | 15 | 54
  Italy | 12 | 5 | 17
  Netherlands | 17 | 6 | 23
  Poland | 64 | 22 | 86
  Romania | 37 | 13 | 50
  Russian Federation | 150 | 55 | 205

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1 (L) at 28 Weeks on Treatment
Description: Trough FEV1 (mean of two highest FEV1 values assessed at 23 and 24 hours after inhalation) at 28 weeks
Time Frame: Week 28
Population: Intention-to-Treat (ITT) population: all randomised patients who took at least one dose of Investigational Medicinal Product and had at least the baseline and one post-baseline value available for the primary efficacy variable.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Aclidinium 200 μg Once-daily: Aclidinium bromide 200 μg once-daily via inhalation
Arm/Group | Aclidinium 200 μg Once-daily | Placebo
Number analyzed (Participants) | 616 | 210
Liters | 1.422 (0.011) | 1.356 (0.017)

2. Secondary Outcome: Time to First Moderate or Severe COPD Exacerbation at 52 Weeks on Treatment
Description: Time to first moderate or severe exacerbation:
  Increase of COPD symptoms during at least 2 consecutive days, treated with antibiotics and/or systemic corticosteroids or an increase in dose of systemic corticosteroids, or leading to hospitalisation.
Time Frame: Week 52
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Aclidinium Bromide 200 μg Once-daily: Aclidinium bromide 200 μg once-daily via inhalation
Arm/Group | Aclidinium Bromide 200 μg Once-daily | Placebo
Number analyzed (Participants) | 616 | 210
Days | NA [NA to NA] — The median time to first moderate or severe COPD exacerbation could not be estimated for either group since fewer than 50% of the population had experienced a moderate or severe exacerbation. | NA [NA to NA] — The median time to first moderate or severe COPD exacerbation could not be estimated for either group since fewer than 50% of the population had experienced a moderate or severe exacerbation.

3. Secondary Outcome: Percentage of Patients Who Achieved at Least a 4-unit Decrease From Baseline in the SGRQ Total Score at 52 Weeks on Treatment
Description: Percentage of patients who achieved a clinically relevant improvement in health-related quality of life at 52 weeks, as measured by at least a 4-unit decrease from baseline in St George's Respiratory Questionnaire (SGRQ) total score
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Aclidinium Bromide 200 μg Once-daily | Placebo
Number analyzed (Participants) | 591 | 200
Percentage of Patients
  Yes (% Patients with 4-unit decrease) | 48.1 | 39.5
  No (% Patients without 4-unit decrease) | 52.0 | 60.5

4. Primary Outcome: Trough Forced Expiratory Volume in the First Second (FEV1) (L) at 12 Weeks on Treatment
Description: Trough FEV1 (mean of two highest FEV1 values assessed at 23 and 24 hours after inhalation) at 12 weeks
Time Frame: Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium 200 μg Once-daily | Placebo
Number analyzed (Participants) | 616 | 210
Liters | 1.428 (0.010) | 1.366 (0.016)

ADVERSE EVENTS:
Time Frame: 52 Weeks
Description: Only COPD exacerbations that were fatal or life-threatening are included here. Other COPD exacerbations were not reported as AEs but were included as part of the efficacy evaluations.
Arm/Group | Aclidinium Bromide 200 μg Once-daily | Placebo
Serious Adverse Events (participants affected / at risk) | 50/627 | 22/216
Other Adverse Events (participants affected / at risk) | 232/627 | 76/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aclidinium Bromide 200 μg Once-daily (N=627) | Placebo (N=216)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Mitrial valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Cataract cortical (Eye disorders) | 1 (1) | 0 (0)
Open angle glaucoma (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 2 (2) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 8 (9) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Phimosis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery emolism (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium Bromide 200 μg Once-daily (N=627) | Placebo (N=216)
Nasopharyngitis (Infections and infestations) | 102 | 31
Headache (Nervous system disorders) | 71 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information related to this clinical trial is considered strictly confidential and is the property of Almirall. This information will not be given to a third party without the written consent of Almirall. Publication and/or presentation, whether complete or partial, of any part of the data or results of this trial will be subject to revision and written agreement between the investigator and Almirall.